CLINICAL TRIAL: NCT05796713
Title: A Quantitative and Qualitative Analysis of the Barriers to Patients' Early Presentation, Diagnosis and Treatment in Childhood Hydrocephalus
Brief Title: Barriers to Patients' Early Presentation, Diagnosis and Treatment in Childhood Hydrocephalus
Status: Completed | Type: Observational
Sponsor: Lagos State University (Other)
Collaborators: Hydrocephalus Association (Other)
Responsible Party: Principal Investigator, Olufemi Idowu, Professor, Lagos State University
Other Study IDs: 2023/Hydro
Record Dates: First submitted 2023-03-07; First posted 2023-04-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hydrocephalus in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hydrocephalus — Interview

SUMMARY:
Patient with childhood hydrocephalus (HC) tend to present late in Low medium income countries (LMICs). This project will study the barriers leading to patients' and health system delay in patients with childhood HC. This will be done via a quantitative and qualitative study analysis. The data will be collected prospectively.

DETAILED DESCRIPTION:
Children less than 5 years of age with HC confirmed with either magnetic resonance or computerized tomographic images will be recruited. In addition, Hospital staff members, who have been working within the Neurosurgical unit for at least 5 years will be interviewed.

The patients' data that will be collected will include gender, age at presentation, socioeconomic class of parents (or guardians), religion, referral source, presenting complaint with its duration, physical findings, ventricular diameter. The Pre-presentation symptoms interval (PPI) will be defined as the number of days between the onset of symptoms and first presentation at any type of healthcare service centre (including primary healthcare centre, secondary health institutions); Presentation Interval (PI)- Number of days from symptoms to presenting at Neurosurgical centre; Pre-diagnostic interval (PDI) will be defined as the interval in days between symptoms and completion of pre-operative investigations. Patient interval (PI) will be defined as the number of days from the onset of symptoms and patient's first contact with the Neurosurgical center. Hospital interval (HI)- number of days from completion of investigations to surgical intervention. The collected data will be analyzed according to qualitative conventional content analysis. Nvivo software version 13 and Statistical Product and Service Solutions (SPSS) version 23 will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients less than 5 years of age with HC confirmed with either magnetic resonance or computerized tomographic images
* Patients' parents' inclusion criteria will be parents (Guardians) of children with radiologically confirmed HC with either magnetic resonance or computerized tomographic images.
* Hospital staff members, who have been working within the Neurosurgical unit for at least 5 years.

Exclusion Criteria:

* All patents not investigated or operated at our centre
* Patients older than 5 years

Max Age: 5 Years | Sex: All
Age Groups: Child
Study Population: Patients who present at the Lagos State University Teaching Hospital, Ikeja, Lagos for management of hydrocephalus
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Patient Presentation time in days | 14 days
  Time in days, from the onset of symptoms to the time the patient seeks medical advice.
Diagnostic delay in days | 14 days
  Time in days between the patient's presentation and the confirmation of the diagnosis, in days
Treatment delay in days | 14 days
  The duration (in days) between the diagnosis and initiation of treatment

SECONDARY OUTCOMES:
Treatment outcome as perceived by parents/caregivers | 4 weeks
  Effectiveness of the treatment in improving patient outcomes using a questionnaire (5-point Likert scale based survey questions with higher scores meaning better outcome)
Parents/caregivers satisfaction | 4 weeks
  The parent's satisfaction with the quality of care received using a questionnaire (5-point Likert scale based survey questions with higher scores meaning better outcome)
Reason for delay in presentation, diagnosis and treatment | 4 weeks
  As described by the parents and hospital staff

CONTACTS AND LOCATIONS:
Overall Officials: Olufemi Idowu, FWACS, FACS, Principal Investigator — Lagos State University Teaching Hospital, Ikeja, Lagos, Nigeria
Locations (1):
- Lagos State University Teaching Hospital, Ikeja, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data on request
Supporting Information: Study Protocol
Time Frame: Jan 2024 till Jan 2025
Access Criteria: via email